CLINICAL TRIAL: NCT03530891
Title: Evaluation of the Efficacy of Computer Guided Lag Screw Fixation in Comparison to Conventional Lag Screw Fixation in Anterior Mandibular Fractures (RCT)
Brief Title: Computer Guided Lag Screw Fixation Versus Conventional Lag Screw Fixation in Anterior Mandibular Fractures
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Cairo University (Other)
Responsible Party: Principal Investigator, Mohamed Kadry, Assistant lecturer, Cairo University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: CEBD-CU-2018-5-4
Record Dates: First submitted 2018-05-04; First posted 2018-05-21 (Actual); Last update posted 2018-05-21 (Actual); Status verified 2018-05

CONDITIONS: Mandible Fracture
Keywords: anterior mandible fracture; surgery computer assisted
MeSH Terms: conditions — Mandibular Fractures | interventions — Surgery, Computer-Assisted

STUDY DESIGN:
Intervention Model Description: * A Randomized clinical trial.
  * Parallel group study.
  * A trial will be carried out in hospital of Oral and Maxillofacial surgery department- Faculty of Oral and Dental Medicine Cairo University
  * Equal randomization: participants with equal probabilities for intervention.
  * Positive controlled: Both groups receiving treatment.
Masking Description: Because the two interventions requires different pre operative preparation, both the participants and investigators can't be blinded.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Computer guided lag screw fixation (Experimental): Patient specific surgical guided will be used for open reduction and internal fixation for anterior mandibular fracture by lag screws.
  Interventions: Procedure: Computer guided lag screw fixation
- Conventional lag screw fixation (Active Comparator): Open reduction and internal fixation for anterior mandibular fracture using lag screws.
  Interventions: Procedure: Conventional lag screw fixation

INTERVENTIONS:
Procedure: Computer guided lag screw fixation — Under general anaesthesia: Patient specific pre operative prefabricated surgical guide will be used intra operative for open reduction and internal fixation for anterior mandibular fracture using lag screws.
  Other Names: computer assisted surgery
  Arms: Computer guided lag screw fixation
Procedure: Conventional lag screw fixation — Under general anaesthesia: Open reduction and internal fixation for anterior mandibular fracture utilising lag screws.
  Other Names: traditional lag screw fixation
  Arms: Conventional lag screw fixation

SUMMARY:
Comparison between computer guided lag screw fixation versus traditional lag screw fixation in open reduction and internal fixation of anterior mandibular fractures.

DETAILED DESCRIPTION:
Two groups of patients with anterior mandibular fractures indicated for open reduction and internal fixation. First group will be subjected to computer guided lag screw fixation. Second group will be subjected to traditional lag screw fixation.

Eligible patients will be randomised in equal proportions between study group (computer guided lag screw fixation) and control group (conventional lag screw fixation).

A- Computer guided lag screw fixation group:

* Pre operative Computed tomography will be done for the patient.
* Computed tomography data will be imported into Computer aided surgical simulation software.
* Utilizing Computer aided surgical simulation software the fracture segments are virtually reduced and patient specific surgical guide is designed and sent to three dimension printer before operation.
* Intra operative: All cases will undergo surgery under general anaesthesia.
* Exposure of the fractured segments will be done using vestibular incision.
* Inter-maxillary fixation will be done
* The fractured segments will be reduced in normal anatomic position guided by occlusion.
* Fracture fragments will be fixed using lag screws utilizing patient specific surgical guide.
* Closure of the surgical incision.
* Post operative at first week Computed tomography will be done for the patient.
* Computed tomography data will be imported into computer aided surgical simulation software.
* Utilizing computer aided surgical simulation software the post operative computed tomography will be superimposed onto the pre operative planned simulation.

B- Conventional titanium plates:

* Pre operative Computed tomography will be done for the patient.
* Computed tomography data will be imported into Computer aided surgical simulation software.
* Utilizing Computer aided surgical simulation software the fracture segments are virtually reduced.
* Intra operative: All cases will undergo surgery under general anaesthesia.
* Exposure of the fractured segments will be done using vestibular incision.
* Inter-maxillary fixation will be done.
* The fractured segments will be reduced in normal anatomic position guided by occlusion.
* The fracture fragments will be fixed using lag screws.
* Closure of the surgical incision.
* Post operative at first week Computed tomography will be done for the patient.
* Computed tomography data will be imported into computer aided surgical simulation software.
* Utilizing computer aided surgical simulation software the post operative computed tomography will be superimposed onto the pre operative planned simulation.

Follow up for both groups:

Clinical evaluation will be performed at first week postoperative then patients will be recalled every week for one month. Final follow up visit will be at 3 months post operative.

ELIGIBILITY:
Inclusion criteria:

* Patients with anterior mandibular fracture indicated for open reduction internal fixation alone or in combination with fracture elsewhere in the mandible or mid face.
* All ages and both sexes were included in this study.
* Patients should be free from any systemic disease that may affect normal healing of bone, and predictable outcome.
* Patients with good general condition allowing major surgical procedure under general anaesthesia .
* Patients with physical and psychological tolerance.

Exclusion criteria:

* Patients with comminuted fractures as it is not indicated for compression osteosynthesis like lag screws.
* Patients with high risk systemic diseases like uncontrolled diabetes mellitus. As uncontrolled diabetes mellitus has a negative impact on normal bone healing.
* Patients with old and/or mal-union fractures. As they will affect accuracy of reduction of the fractured segments.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 26 (Estimated)
Dates: Start 2018-01-11 (Actual); Primary Completion 2019-03-01 (Estimated); Study Completion 2019-06-01 (Estimated)

PRIMARY OUTCOMES:
Stability of fixed fractured segment | 1st week post operative.
  stability of fixed fractured segment will be assessed using measuring device bimanual manipulation, measuring unit (binary yes or no)

SECONDARY OUTCOMES:
neurosensory disturbance | one month post operative
  presence of neurosensory disturbance will be assessed using measuring device: subjective assessment, measuring unit (binary yes or no)
Accuracy of lag screw placement | 1st week post operative.
  Accuracy of lag screw placement will be assessed by measuring device: Computer aided surgical simulation (CASS) software, measuring unit: Millimetre
supplemental fixation devices | intra operative and one month post operative
  The need for intra operative or post operative supplemental fixation devices, measuring device clinical assessment. measuring unit: binary yes or no
Need for second surgery | one month post operative
  The need for second surgical procedure will be assessed by clinical assessment (measuring device). measuring unit: binary (yes or no).

CONTACTS AND LOCATIONS:
Overall Officials: Khaled S Amr, PhD, Study Director — Faculty of oral and dental medicine, Cairo University.
Locations (1):
- Faculty of Oral and Dental Medicine - Cairo University, Giza, Egypt

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Ellis E 3rd, Ghali GE. Lag screw fixation of anterior mandibular fractures. J Oral Maxillofac Surg. 1991 Jan;49(1):13-21; discussion 21-2. doi: 10.1016/0278-2391(91)90259-o. PMID 1985177
- [Background] Ellis E 3rd. Is lag screw fixation superior to plate fixation to treat fractures of the mandibular symphysis? J Oral Maxillofac Surg. 2012 Apr;70(4):875-82. doi: 10.1016/j.joms.2011.08.042. Epub 2011 Dec 30. PMID 22209100
- [Background] Kallela I, Ilzuka T, Laine P, Lindqvist C. Lag-screw fixation of mandibular parasymphyseal and angle fractures. Oral Surg Oral Med Oral Pathol Oral Radiol Endod. 1996 Nov;82(5):510-6. doi: 10.1016/s1079-2104(96)80195-8. PMID 8936514
- [Background] Xia JJ, Gateno J, Teichgraeber JF, Christensen AM, Lasky RE, Lemoine JJ, Liebschner MA. Accuracy of the computer-aided surgical simulation (CASS) system in the treatment of patients with complex craniomaxillofacial deformity: A pilot study. J Oral Maxillofac Surg. 2007 Feb;65(2):248-54. doi: 10.1016/j.joms.2006.10.005. PMID 17236929
- [Background] Zachariades N, Mezitis M, Papademetriou I. Use of lag screws for the management of mandibular trauma. Oral Surg Oral Med Oral Pathol Oral Radiol Endod. 1996 Feb;81(2):164-7. doi: 10.1016/s1079-2104(96)80407-0. PMID 8665308
- [Background] Tiwana PS, Kushner GM, Alpert B. Lag screw fixation of anterior mandibular fractures: a retrospective analysis of intraoperative and postoperative complications. J Oral Maxillofac Surg. 2007 Jun;65(6):1180-5. doi: 10.1016/j.joms.2006.11.046. PMID 17517303
- [Background] Jones JK, Van Sickels JE. Rigid fixation: a review of concepts and treatment of fractures. Oral Surg Oral Med Oral Pathol. 1988 Jan;65(1):13-8. doi: 10.1016/0030-4220(88)90183-1. PMID 3277107
- [Background] Retzepi M, Donos N. The effect of diabetes mellitus on osseous healing. Clin Oral Implants Res. 2010 Jul;21(7):673-81. doi: 10.1111/j.1600-0501.2010.01923.x. Epub 2010 May 3. PMID 20465554
- [Background] Parashar A, Sharma RK. Unfavourable outcomes in maxillofacial injuries: How to avoid and manage. Indian J Plast Surg. 2013 May;46(2):221-34. doi: 10.4103/0970-0358.118597. PMID 24501458